CLINICAL TRIAL: NCT07129434
Title: Strengthening Healthy Emotional Co-regulation of Mothers With PCOS and Obesity and Their Infants
Acronym: ECoFam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Principal Investigator, Julia Jaekel, Prof. Dr., Oulu University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ECoFam PEPPI Pilot RCT
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Obesity &Amp;Amp; Overweight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Overweight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECoFam intervention (Experimental): personalized coaching sessions
  Interventions: Behavioral: ECoFam
- treatment-as-usual (TAU) (No Intervention): control group, no intervention administered

INTERVENTIONS:
Behavioral: ECoFam — Mother-infant dyads randomized into the intervention group receive four personal coaching sessions to facilitate emotional connection via multisensory channels including comfort touch and communication of face-to-face affect during holding time.
  Arms: ECoFam intervention

SUMMARY:
It is both timely and important to invest in interventions that can improve healthy emotional co-regulation. It is proposed to evaluate the feasibility and limited efficacy of an adapted, brief, multimodal intervention: ECoFam (Emotional connection and Co-regulation for Families). Evidence from the US suggests intervention effects on maternal and infant outcomes that are large in effect size (i.e., Cohen's d >0.6 for increasing emotional connection and decreasing maternal depressive symptoms) (21-23). The study results will directly translate evidence into practice and, if found feasible, allow rapid scaling-up.

Objectives:

1. Build capacity for implementation of a novel diagnostic screening tool for emotional co-regulation, the uWECS, as part of clinical follow-up for mother-infant dyads with high fibrobesity risk in Finland.
2. Test the feasibility and limited efficacy of the brief, multimodal ECoFam intervention to foster healthy emotional co-regulation between mothers with PCOS and obesity and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS
* Obesity according to BMI
* Gave birth at Oulu University Hospital in 2024-25
* PEPPI cohort study participation
* uWECS emotional connection score <9.0 at pre-test

Exclusion Criteria:

- Infant death

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Universal Welch Emotional Connection Screen (uWECS) | From enrollment to the end of intervention and follow-up at 4 months
  Emotional connection evaluated with the uWECS

SECONDARY OUTCOMES:
Mothers' mental health problems | From enrollment to end of intervention and follow-up 4 months
  Mothers' mental health problems are assessed with a range of standardized questionnaires using RedCap; higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Jäkel, Dr. phil. habil., Principal Investigator — University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No